CLINICAL TRIAL: NCT06084663
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Oral Dose, Cross Over Bioequivalence Study of Two Products of Apremilast 30 mg Tablets in Normal, Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Two Products of Apremilast 30 mg Tablets in Healthy, Adult, Human Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0005-22
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Psoriasis and Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apremilast 30 mg Tablets (Experimental): One tablet was administered orally to each subject as per randomization schedule in each period
  Interventions: Drug: Apremilast 30 mg Tablets; Drug: Otezla 30 mg film-coated tablets
- Otezla 30 mg film-coated tablets (Active Comparator): One tablet was administered orally to each subject as per randomization schedule in each period
  Interventions: Drug: Apremilast 30 mg Tablets; Drug: Otezla 30 mg film-coated tablets

INTERVENTIONS:
Drug: Apremilast 30 mg Tablets — Each film-coated tablet contains 30 mg of apremilast
Drug: Otezla 30 mg film-coated tablets — Each film-coated tablet contains 30 mg of apremilast

SUMMARY:
An open label, balanced, randomized, two-sequence, two-treatment, two-period, single oral dose, crossover, bioequivalence study in normal, healthy, adult, human subjects under fasting condition

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker, Normal, healthy, adult, human, subjects between 18 and 45 years of age (both inclusive).
* Having a Body Mass Index (BMI) between 18.5 to 30.0 (both inclusive), calculated as weight in kg/height in m2.
* Not having significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12 lead ECG, and chest X-ray recordings (P/A view).
* Able to understand and comply with the study procedures, in the opinion of the investigator.
* Able to give voluntary written informed consent for participation in the trial.
* In case of female subjects:

Surgically sterilized at least 6 months prior to study participation. Or If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And Serum pregnancy test must be negative.

Exclusion Criteria:

* History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion or Use of medication [non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines)] at any time from 14 days prior to dosing of period-I and Use of any prescribed systemic or topical medication from 30 days prior to dosing of period-I and any vaccine (including COVID-19 vaccine) within 14 days prior to dosing of period-I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
* Consumption of grapefruits or its products within a period of 72 hours prior to dosing of period-I.
* Smokers or who have smoked within last 06 months prior to start of the study.
* A recent history of harmful use of alcohol (less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to dosing of period-I.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre study drug scans.
* History or presence of seizure or psychiatric disorder
* A history of difficulty with donating blood.
* Donation of blood (1 unit or 350 mL) within a period of 90 days prior to the first dose of study medication.
* Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication**.
* ** If investigational medicinal product is received within 90 days where there is no blood loss except safety lab testing, subject can be included considering 10 half-lives duration of investigational medicinal product received.
* Difficulty in swallowing tablet or oral solid dosage form
* A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.
* A positive test result for HIV antibody (1 &/or 2).
* An unusual diet, for whatever reason (for example, fasting, high potassium or low-sodium), for four weeks prior to receiving the study drug in period I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Any condition which places the subject at unacceptable risk if he/she were to participate in the study, or confounds the ability to interpret data from the study.
* Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure, colon resection, irritable bowel syndrome, Crohn's disease, etc.
* The QTc interval more than 450 msec for male subjects and 460 msec for female subjects at the time of screening.
* Nursing mothers (for female subjects).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Cmax | The venous blood samples will be withdrawn at pre-dose (0.000 hour) and at 0.250, 0.500, 0.750, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 5.000, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000 and 48.000 hours
  Maximum plasma concentration
AUC0-t | The venous blood samples will be withdrawn at pre-dose (0.000 hour) and at 0.250, 0.500, 0.750, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 5.000, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000 and 48.000 hours
  Area under the plasma concentration curve from administration to last observed concentration at time t

SECONDARY OUTCOMES:
AUC0-∞ | The venous blood samples will be withdrawn at pre-dose (0.000 hour) and at 0.250, 0.500, 0.750, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 5.000, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000 and 48.000 hours
  Area under the plasma concentration curve extrapolated to infinite time

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No